CLINICAL TRIAL: NCT02817802
Title: BIOTRONIKS - Safety and Performance in de NOvo Lesion of NatiVE Coronary Arteries With Magmaris- Registry: BIOSOLVE-IV
Acronym: BIOSOLVE-IV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C1503
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Coronary Artery Disease
Keywords: Registry; Magmaris; Coronary Artery Disease; PCI
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Magmaris: Magmaris Sirolimus-Eluting Resorbable Coronary Magnesium Scaffold
  Interventions: Device: Magmaris

INTERVENTIONS:
Device: Magmaris — PCI (Magmaris)

SUMMARY:
The registry will investigate the clinical performance and long-term safety of Magmaris in a real world setting

DETAILED DESCRIPTION:
Coronary stents are the default devices for the treatment of coronary artery disease in percutaneous coronary intervention (PCI) according to existing guidelines. However, thrombosis and restenosis are still the main limitations of current permanent metallic stents. In contrast to Bare Metal Stents (BMSs), Drug Eluting Stents (DESs) have a reduced restenosis rate due to the presence of antiproliferative agents in the coating layer of the stent surface and reduced rate of repeat revascularisation. However, late and very late stent thrombosis remains the limitation of DES in spite of prolonged dual antiplatelet therapy.Bioabsorbable scaffolds have been introduced to overcome limitations of permanent metallic stents.

The aim of this observational registry is to investigate the clinical performance and long-term safety of Magmaris in a real world setting.

ELIGIBILITY:
Inclusion cirteria

1. Subject is ≥18 years of Age
2. Subject must be willing to sign a Patient Informed Consent (PIC) or Patient Data Release Form (PDRF) where applicable
3. Symptomatic coronary artery disease
4. Subject with a maximum of two single de novo lesions in two different major epicardial vessels
5. Target lesion length ≤21 mm by QCA or by visual estimation
6. Target lesion stenosis by visual estimation: >50% - <100% and TIMI flow ≥1
7. Subject is eligible for Dual Anti Platelet Therapy (DAPT)
8. Reference vessel diameter between 2.7-3.7 mm by visual estimation, depending on the scaffold size used

Exclusion criteria

1. Pregnant and/or breast feeding females or females who intend to become pregnant during the time of the registry
2. Known allergies to: Acetylsalicylic Acid (ASA), clopidogrel, ticlopidin, heparin or any other anticoagulant/antiplatelet required for PCI, contrast medium, sirolimus, or similar drugs; or the scaffold materials including Magnesium, Yttrium, Neodymium, Zirconium,Gadolinium, Dysprosium, Tantalum that cannot beadequately pre-medicated
3. Subjects on dialysis
4. Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute ST Elevation myocardial infarction (STEMI) within 72 hours prior to the index procedure. Note: Hemodynamically stable non-STEMI (NSTEMI) subjects are eligible for study enrollment
5. Documented left ventricular ejection fraction (LVEF) <30%
6. Restenotic target lesion
7. Thrombus in target vessel
8. Target lesion is located in or supplied by a diseased (defined as vessel irregularity per angiogram and >20% stenosed lesion by visual estimation) arterial or venous bypass graft
9. Left main coronary artery disease
10. Ostial target lesion (within 5.0 mm of vessel origin)
11. Target lesion involves a side branch ≥2.0 mm in Diameter
12. Target vessel (including side branches) has second lesion which requires treatment according to the investigator's discretion
13. Unsuccessful pre-dilatation, defined as residual Stenosis rate more than 20% measured by QCA and / or angiographic complications (e.g. distal embolization, side branch closure, extensive dissections)
14. Planned surgery within 6 months of PCI unless dual antiplatelet therapy will be maintained
15. Currently participating in another study and Primary endpoint is not reached yet.
16. Planned interventional treatment of any target or nontarget vessel

Participating Countries

Australia, Austria, Belgium, Denmark, France, Germany, Hong Kong, Hungary, Israel, Italy, Latvia, Malaysia, New Zealand, Poland, Portugal, Singapore, South Africa, South Korea, Spain, Sweden, Switzerland, Taiwan, Thailand, The Netherlands, United Kingdom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic coronary artery disease needing the treatment of de novo native coronary artery lesions.
Sampling Method: Non-Probability Sample
Enrollment: 2066 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF)* at 12 months | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Verheye, MD, Principal Investigator — Cardiovascular Institute Middelheim, Antwerpen, Belgium; Michael Kang-Yin Lee, MD, Principal Investigator — Queen Elizabeth Hospital, Hong Kong
Locations (2):
- ZNA Middelheim Cardiologiy, Antwerp, Belgium
- Queen Elizabeth Hospital, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The primary outcome data will be shared after the publication of it.

REFERENCES:
- See also: Primary end point of the study — https://pubmed.ncbi.nlm.nih.gov/32881396/